CLINICAL TRIAL: NCT07234344
Title: A Predictive Model for Midwives' Compassion Fatigue: A Cross-Sectional Study
Brief Title: A Predictive Model for Midwives' C F: A Cross-Sectional Study
Status: Completed | Type: Observational
Sponsor: LanZhou University (Other)
Responsible Party: Principal Investigator, Zhan Yian, student, LanZhou University
Other Study IDs: LZUHLXY20250053
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Compassion Fatigue
MeSH Terms: conditions — Compassion Fatigue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Compassion fatigue is a professional psychological problem caused by long-term work pressure, resulting in emotional exhaustion and a decline in empathy ability. It not only leads to individual symptoms such as sleep disorders and anxiety, but also increases clinical errors, reduces work efficiency, and causes the loss of medical talents. It has become a common challenge faced by medical staff worldwide. In the international medical system, midwives, as the core force safeguarding the health of mothers and infants, are working in an increasingly complex and high-pressure environment. Midwives, due to their continuous engagement of a large amount of emotional labor and frequent exposure to multiple pressures such as traumatic events during childbirth, obstetric emergency complications, and occupational exposure, have become a high-risk group for compassion fatigue.

The causes of compassion fatigue among midwives are complex and diverse. Moreover, most of the existing assessment tools for compassion fatigue are universal assessment scales, and the unique risks of midwives' work have not yet been highlighted and reflected. Therefore, it is urgent to establish an compassion fatigue assessment tool specifically for the midwife population, so as to accurately and efficiently identify the compassion fatigue status of midwives, provide a reference for managers to grasp the current situation of compassion fatigue among midwives, and formulate efficient and targeted management and take corresponding intervention measures, thereby effectively reducing the incidence of empathy fatigue among midwives.

This study summarized the factors that may affect the occurrence of compassion fatigue among midwives through literature review and clinical practice, conducted a cross-sectional study to explore the influencing factors of compassion fatigue among midwives, and established a nomogram prediction model, with the aim of helping clinical managers simply and quickly screen out high-risk groups of compassion fatigue It provides a reference basis for taking targeted and preventive management measures at an early stage.

ELIGIBILITY:
Inclusion Criteria:

* Possession of a midwifery practice license; currently engaged in midwifery practice; midwifery practice duration > 1 year; voluntary participation in the study, and signed informed consent.

Exclusion Criteria:

* History of psychiatric disorders; use of psychiatric medications within one month before the survey.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Within the international healthcare system, midwives serve as a core force safeguarding maternal and infant health, yet their working environment is becoming increasingly complex and high-pressure. Due to their sustained investment of significant emotional labor and frequent exposure to multiple stressors-including traumatic events during childbirth, obstetric emergencies, and occupational exposures-midwives have become a high-risk group for compassion fatigue .
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2025-09-16 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
compassion fatigue | September 16 to 30, 2025
  The Professional Quality of Life Scale was developed by Stamm et al. in 2005 to measure compassion fatigue among research subjects. In 2013, Chinese scholar Chen Huaying translated, adapted, and revised the original scale to create the Chinese version of the Compassion Fatigue Scale, incorporating Chinese cultural contexts and national conditions . The scale comprises 30 items across three dimensions: Empathic Satisfaction, Burnout, and Secondary Traumatic Stress, with 10 items per dimension. Items are rated on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). This scale demonstrates good reliability and validity among Chinese clinical nurses, with a Cronbach's α coefficient of 0.91. The Cronbach's α coefficients for the three dimensions are 0.87, 0.73, and 0.84, respectively. It is suitable for assessing compassion fatigue levels among midwives.

SECONDARY OUTCOMES:
Midwife Trauma Stress | September 16 to 30, 2025
  The Midwife Trauma Stress Scale was developed by Kubota et al. in 2022 to measure the frequency and impact of traumatic stress events experienced by midwives. Due to differences in healthcare environments and cultures, Chinese researchers Pu adapted it cross-culturally by removing Item 12 and modifying certain phrasing to enhance readability for study participants . This unidimensional scale comprises 15 items organized into two subscales: occurrence frequency and impact severity. Each item uses a 4-point Likert scale. Scores of 0-3 for occurrence frequency and impact severity correspond to 'never occurred' to 'frequently occurred' and 'no impact' to 'significant impact,' respectively. The scale does not calculate a total score. Both subscales range from 0 to 45 points, with higher scores indicating greater frequency of traumatic stress events experienced by midwives and more severe physical and psychological impact.
Social Support | September 16 to 30, 2025
  The Social Support Scale was developed by Xiao Shuiyuan in 1986 to measure the degree of social support received by individuals. The scale comprises 10 items across three dimensions: objective support, subjective support, and utilization of support. Item 5 is subdivided into four sections (A, B, C, D) for total scoring, with each section rated from 1 (none) to 4 (full support); Items 6 and 7 assign 0 points for 'no sources' and corresponding points for 'specific sources' based on the number selected, ranging from 0 to 9 points. Other items assign 1, 2, 3, or 4 points for selecting 1, 2, 3, or 4 options, respectively. A total scale score <33 indicates low social support, 33-45 indicates moderate social support, and >45 indicates high social support. Higher total scores reflect greater social support.
Psychological Resilience | September 16 to 30, 2025
  The 10-item Connor-Davidson Resilience Scale was revised by Campbell-Sills et al. based on the 25-item Connor-Davidson Resilience Scale (CD-RISC) developed by Connor et al. in 2003. Chinese researchers Wang Li et al. adapted it through cross-cultural adjustments and reliability/validity testing to create the Simplified Psychological Resilience Scale. This 10-item scale employs a 5-point Likert scale, with responses ranging from 0 (almost never) to 4 (always). Total scores range from 0 to 40, with higher scores indicating greater psychological resilience. The scale demonstrated a Cronbach's α coefficient of 0.91 and a test-retest reliability coefficient of 0.90. It has shown good reliability and validity across multiple studies and is suitable for assessing midwives' psychological resilience levels.
simplified coping style | September 16 to 30, 2025
  The Simplified Coping Strategies Questionnaire, developed by Xie Yaning in 1998 based on a synthesis of relevant coping theory, assesses the attitudes and approaches research subjects may adopt when facing setbacks or difficulties. This 20-item scale comprises two dimensions: positive coping (12 items) and negative coping (8 items). It employs a 4-point Likert scale: 0, 1, 2, and 3 represent 'never,' 'rarely,' 'sometimes,' and 'often,' respectively. A coping tendency score greater than 0 indicates the respondent primarily uses positive coping strategies under stress, while a score less than 0 suggests a tendency toward negative coping strategies.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, Lanzhou Universit, Lanzhou City, Gansu, Gansu, China